CLINICAL TRIAL: NCT01397474
Title: Peripheral Perfusion Targeted Fluid Management in Critically Ill Patients: a Pilot Study
Brief Title: Peripheral Perfusion Targeted Fluid Management
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, ME van Genderen, Drs, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NL34607.078.10
Record Dates: First submitted 2011-07-07; First posted 2011-07-19 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Sepsis; Severe Sepsis
Keywords: peripheral perfusion; critically ill patients; fluid administration
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): The fluid management algorithm of the control group is based on the standard care procedure of our ICU as recommended in guidelines: the patient's fluid status is assessed by performing a fluid challenge with a bolus of 250 ml colloids. When the patients is fluid responsive (i.e. showing an increase in stroke volume > 10% ) he will receive an additional bolus of 250 ml of colloids. After each fluid challenge, patients will be revaluated for fluid responsiveness to access need of further fluid administration.
- PPTFM (Experimental): The fluid management algorithm of the intervention group uses identical therapy (i.e. fluids) yet targeted at different endpoints (i.e. peripheral perfusion parameters). After evaluation of peripheral perfusion, only patients with a "bad peripheral perfusion" (i.e. 3 out of 4 criteria considered as bad) will receive a fluid challenge, the same way as in the standard care procedure (i.e. bolus of 250 ml of fluid). After each fluid challenge, patients will be re-evaluated for peripheral perfusion to access further need in fluid challenges. To ensure that no hypovolemia will occur in the intervention group, fluid will be administered irrespectively of peripheral perfusion parameters, if cardiac index falls below a value of 2,5 L/min/m2.
  Interventions: Other: PPTFM

INTERVENTIONS:
Other: PPTFM — Peripheral Perfusion Targeted Fluid Management
  Other Names: CRT; PFI; delta Temp; StO2
  Arms: PPTFM

SUMMARY:
* Impaired peripheral perfusion is related to worse outcome in critically ill patients. Although this is known, these parameters have never been used as target for hemodynamic therapy.
* We hypothesize that targeting of fluid administration on parameters of peripheral perfusion might prevent excessive fluid administration, leading to less formation of tissue edema, less respiratory dysfunction and shorter duration of mechanical ventilation in critically ill patients.

DETAILED DESCRIPTION:
Rationale: Currently, fluid administration of critically ill patients is aimed at optimizing conventional hemodynamic parameters such as stroke volume and cardiac output. Fluid is infused repeatedly until patients become "non-responsive", i.e. cardiac output does not increase anymore. However, the ultimate goal of hemodynamic therapy should be to improve peripheral (i.e. tissue) perfusion. Recently we have shown that 1) increasing stroke volume does not always have an effect on peripheral perfusion and 2) that peripheral perfusion is not impaired when stroke volume can still be increased with fluid infusion. Furthermore, repeated administration of fluid in order to reach a maximum cardiac output can lead to an enormous accumulation of fluid in the patient. This leads to formation of lung edema and respiratory dysfunction and is associated with prolonged mechanical ventilation and ICU-stay. Recently, techniques have been developed which allow bedside assessment of peripheral perfusion. Although impaired peripheral perfusion was related to worse outcome, these parameters have never been used as target for hemodynamic therapy.

Objective: To study whether peripheral perfusion targeted fluid management (PPTFM) leads to less fluid administration, improved respiratory function and shorter mechanical ventilation.

Study design: The study is a pilot study and is designed as a randomized controlled trial. The study will be conducted as a single-center study at the Intensive Care of the Erasmus Medical Center.

Study population: We aim to include 40 adult patients who are admitted to the Intensive Care with hemodynamic instability (defined as mean arterial pressure < 65 mmHg and an arterial lactate concentration > 3.0 mmol/l) due to severe sepsis and septic shock.

Intervention: In the intervention group fluid management is targeted on peripheral perfusion parameters while in the control group fluid is administered in order to optimize cardiac output.

Main study parameters/endpoints: The main study endpoints are daily fluid balance and duration of mechanical ventilation.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There is a possible risk that in the treatment group the patients will remain hypovolemic. To ensure that this will not occur, fluids will be administrated in this group, irrespective of peripheral perfusion parameters, until cardiac index is 2,5 L/min/m2. Assessment of peripheral perfusion is performed with non-invasive optical techniques that impose no burden to the patient.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (>18 years) admitted to the intensive care with 1) hemodynamic instability due to severe sepsis, and 2) a mean arterial pressure < 65 mmHg and 3) an arterial lactate concentration > 3.0 mmol/L will be considered for participation

Exclusion Criteria:

* moribund.
* severe coagulation disorder (contraindication for central venous catheter placement).
* severe peripheral vascular disease (interfering with peripheral perfusion measurement).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Fluid balance during Intensive Care Unit stay | untill 72 hours after admission
  Total and daily fuid balance for a maximal time period of 72 hours

SECONDARY OUTCOMES:
CRT (Capillary refill time) | Within 72 hours after admission
  Parameter of peripheral perfusion
Systemic hemodynamic variables | Untill 72 hours after admission to the ICU
  * Heart Rate
  * Mean Arterial Pressure
  * Cardiac Index
  * Cardiac output
  * Stroke Volume
  * Central Venous Pressure
  * Systemic Vascular Resistance
Respiratory function | Untill 72 hours after admission to the ICU
  * FiO2
  * PEEP
  * Breathing Frequency
  * pCO2
  * pO2
PFI (Peripheral Flow Index) | Untill 72 hours after ICU admission
  Parameter of peripheral perfusion
Tskindiff (Forearm-to-Fingertip temperature skin difference) | Untill 72 hours after ICU admission
  Parameter of peripheral perfusion
StO2 (Peripheral tissue oxygenation) | Untill 72 hours after ICU admission
  Parameter of peripheral perfusion

CONTACTS AND LOCATIONS:
Overall Officials: Jasper van Bommel, MD, PhD, Study Director — Erasmus Medical Center; Michel E Genderen, Drs, Principal Investigator — Erasmus Medical Center
Locations (1):
- ErasmusMC, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Background] Lima A, Jansen TC, van Bommel J, Ince C, Bakker J. The prognostic value of the subjective assessment of peripheral perfusion in critically ill patients. Crit Care Med. 2009 Mar;37(3):934-8. doi: 10.1097/CCM.0b013e31819869db. PMID 19237899
- [Background] Lima A, van Bommel J, Sikorska K, van Genderen M, Klijn E, Lesaffre E, Ince C, Bakker J. The relation of near-infrared spectroscopy with changes in peripheral circulation in critically ill patients. Crit Care Med. 2011 Jul;39(7):1649-54. doi: 10.1097/CCM.0b013e3182186675. PMID 21685739
- [Derived] van Genderen ME, Engels N, van der Valk RJ, Lima A, Klijn E, Bakker J, van Bommel J. Early peripheral perfusion-guided fluid therapy in patients with septic shock. Am J Respir Crit Care Med. 2015 Feb 15;191(4):477-80. doi: 10.1164/rccm.201408-1575LE. No abstract available. PMID 25679107